CLINICAL TRIAL: NCT00283387
Title: Efficacy of Betaine for Reduction of Urine Oxalate in Patients With Type 1 Primary Hyperoxaluria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Orphan Europe (Unknown)
Responsible Party: Dr. Carla G. Monico, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2147-05; 5R01DK073354-04 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Hyperoxaluria
Keywords: Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria; Hyperoxaluria, Primary | interventions — Betaine; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betaine (Experimental): Subjects were randomly assigned oral betaine 12 grams/day in subjects younger than 10 years of age, and 20 grams/day in subjects 10 years of age and older, in two divided doses. This was followed by a 2 month washout period. Subjects then received the alternative study medication, oral lactose placebo, in two doses daily, for 2 months.
  Interventions: Drug: Betaine; Drug: Placebo
- Placebo (Placebo Comparator): Subjects were randomly assigned to receive oral lactose placebo, in two doses daily, for 2 months. This was followed by a 2 month washout period. Subjects then received the alternative study medication, oral betaine 12 grams/day in subjects younger than 10 years of age, and 20 grams/day in subjects 10 years of age and older, in two divided doses, for 2 months.
  Interventions: Drug: Betaine; Drug: Placebo

INTERVENTIONS:
Drug: Betaine — Subjects were randomly assigned oral betaine 12 grams/day in subjects younger than 10 years of age, and 20 grams/day in subjects 10 years of age and older, in two divided doses, for 2 months.
  Other Names: Cystadane
Drug: Placebo — Subjects received oral lactose placebo, in two doses daily, for 2 months.
  Other Names: Lactose

SUMMARY:
The aim of this study is to assess the efficacy and safety of betaine in reducing urine oxalate excretion of Type 1 Primary Hyperoxaluria (PHI) patients.

Hypothesis:

Betaine will effectively reduce urine oxalate excretion in Primary Hyperoxaluria Type I patients.

DETAILED DESCRIPTION:
Our prior genotyping results have shown an association between the G170R allele and the clinical response to VB6. Patients homozygous for this change show a complete response and heterozygous patients a partial response. Since VB6 is a safe and completely effective treatment for patients homozygous for G170R, we will not study betaine in this group. Instead, 20 participants older than 6 years of age who are G170R compound heterozygous, non-G170R missense or truncating sequence change homozygous or heterozygous, will be selected for enrollment. Participants in whom VB6 provides a partial reduction in urine oxalate excretion (compound heterozygotes for the G170R mutation) will be maintained on a stable dose of VB6 (8 mg/kg/d) for two months before and throughout betaine treatment. Those who have demonstrated no response to VB6 will receive betaine alone.

Participants will be randomized to receive either betaine or placebo for the first 2 month arm of the study. Following 2 months of treatment and 2 months of washout, each participant will cross over to the other arm of the study. The other arm will consist of the participant being on 2 months of treatment of whatever they were not taking in the first arm (betaine vs. placebo). Neither the study staff nor the participant will know whether the participant is taking betaine for the first or second arm of the study, or the placebo for the first or second arm of the study. Only the pharmacy will know this.

Prior to the study, a complete history and physical examination, and baseline laboratory studies pertinent to the routine care of primary hyperoxaluria patients will be performed (Complete Blood Count (CBC) with differential, chemistry group, electrolytes, plasma oxalate and creatinine clearance, urinary supersaturation). All women capable of reproduction will receive a pregnancy test prior to enrollment.

Participant will complete two 24-hour urine collections for calcium oxalate super-saturation (includes 24-hour urine oxalate excretion) at baseline, inclusive of creatinine determination for assessment of completeness. They will then begin Cystadane anhydrous solution (12 grams/day in subjects younger than 10 years of age, and 20 grams/day in subjects 10 years of age and older, in two divided doses). These doses of betaine have been shown to effectively treat pediatric patients with VB6-resistant homocystinuria and reverse Nonalcoholic Steatohepatitis (NASH) in adult patients, so we expect they will achieve sufficient intra-hepatocyte levels to have an effect in PHI.

A sample of each 24-hour urine will be stored frozen (-80ºC) to allow determination of indicators of oxidant stress, should urinary oxalate fall.

If effective, betaine could represent a new and safe treatment option for a subset of PHI patients, particularly those with either partially VB6 responsive or VB6 refractory hyperoxaluria, or those with adverse effects such as peripheral neuropathy from large doses of VB6. We do not anticipate any adverse medication effects specific to primary hyperoxaluria. However, as an extra safeguard for children with PHI, ten subjects older than 15 years of age will be tested first and if the agent is well tolerated in PHI patients, pediatric subjects older than 6 years of age will then be recruited for participation.

ELIGIBILITY:
Inclusion Criteria:

1. A definitive diagnosis of Type 1 Primary Hyperoxaluria (PHI) as confirmed by hepatic angiotensinogen (AGT) deficiency, biochemical criteria (marked hyperoxaluria and hyperglycolic aciduria) or mutation analysis (having a known PHI mutation)
2. Alanine-glyoxylate aminotransferase (AGXT) genotype known
3. Hyperoxaluria not fully corrected by 3 months of continuous Vitamin B6 (VB6) at doses of 8 mg/kg/d or more
4. Males or females, 6-70 years of age, inclusive
5. Preserved renal function, as defined by measured glomerular filtration rate (GFR) > 30 ml/min/1.73 m^2
6. Sexually active female patients of childbearing potential must practice adequate contraception during the treatment period and for 6 months after discontinuation of therapy. A pregnancy test obtained at entry prior to the initiation of treatment must be negative. Female patients must not be breast-feeding. Sexually active male patients must practice acceptable methods of contraception during the treatment period and for 6 months after discontinuation of therapy.
7. Written informed consent for participation in this study.

Exclusion Criteria:

1. Patients who are fully VB6 responsive (i.e., G170R homozygotes).
2. Prior recipients of liver transplantation performed for correction of AGT deficiency.
3. Pregnancy or breastfeeding
4. Unwillingness of patient and/or partner to use contraception during treatment.
5. Malignant disease (other than non-melanoma skin cancer) in the previous two years.
6. Markedly reduced renal function (Stage IV Chronic Kidney Disease or measured or estimated GFR < 30 ml/min/1.73 m^2)
7. Allergy to betaine or related compounds
8. History of papilledema or increased intracranial pressure.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla G Monico, M.D., Principal Investigator — Mayo Clinic Hyperoxaluria Center, Rochester MN
Locations (1):
- Mayo Clinic Hyperoxaluria Center, Rochester, Minnesota, United States

REFERENCES:
- [Background] Abdelmalek MF, Angulo P, Jorgensen RA, Sylvestre PB, Lindor KD. Betaine, a promising new agent for patients with nonalcoholic steatohepatitis: results of a pilot study. Am J Gastroenterol. 2001 Sep;96(9):2711-7. doi: 10.1111/j.1572-0241.2001.04129.x. PMID 11569700
- [Background] Adamzik M, Schmermund A, Reed JE, Adamzik S, Behrenbeck T, Sheedy PF 2nd. Comparison of two different software systems for electron-beam CT-derived quantification of coronary calcification. Invest Radiol. 1999 Dec;34(12):767-73. doi: 10.1097/00004424-199912000-00006. PMID 10587873
- [Background] ARCHER HE, DORMER AE, SCOWEN EF, WATTS RW. Primary hyperoxaluria. Lancet. 1957 Aug 17;273(6990):320-2. doi: 10.1016/s0140-6736(57)92210-9. No abstract available. PMID 13464052
- [Background] Barak AJ, Beckenhauer HC, Badakhsh S, Tuma DJ. The effect of betaine in reversing alcoholic steatosis. Alcohol Clin Exp Res. 1997 Sep;21(6):1100-2. PMID 9309323
- [Background] Bourot S, Sire O, Trautwetter A, Touze T, Wu LF, Blanco C, Bernard T. Glycine betaine-assisted protein folding in a lysA mutant of Escherichia coli. J Biol Chem. 2000 Jan 14;275(2):1050-6. doi: 10.1074/jbc.275.2.1050. PMID 10625645
- [Background] Cochat P, Deloraine A, Rotily M, Olive F, Liponski I, Deries N. Epidemiology of primary hyperoxaluria type 1. Societe de Nephrologie and the Societe de Nephrologie Pediatrique. Nephrol Dial Transplant. 1995;10 Suppl 8:3-7. doi: 10.1093/ndt/10.supp8.3. PMID 8592622
- [Background] Danpure CJ and Rumsby G. Enzymology and molecular genetics of primary hyperoxaluria type 1. Consequences for clinical management. In: Calcium Oxalate in Biological Systems, edited by Khan SR. Boca Raton, FL: CRC Press, 1995, p. 189-205.
- [Background] Diamant S, Eliahu N, Rosenthal D, Goloubinoff P. Chemical chaperones regulate molecular chaperones in vitro and in cells under combined salt and heat stresses. J Biol Chem. 2001 Oct 26;276(43):39586-91. doi: 10.1074/jbc.M103081200. Epub 2001 Aug 21. PMID 11517217
- [Background] Diamant S, Rosenthal D, Azem A, Eliahu N, Ben-Zvi AP, Goloubinoff P. Dicarboxylic amino acids and glycine-betaine regulate chaperone-mediated protein-disaggregation under stress. Mol Microbiol. 2003 Jul;49(2):401-10. doi: 10.1046/j.1365-2958.2003.03553.x. PMID 12828638
- [Background] Levine DZ, Nash LA, Chan T, Dubrovskis AH. Proximal bicarbonate reabsorption during Ringer and albumin infusions in the rat. J Clin Invest. 1976 Jun;57(6):1490-7. doi: 10.1172/JCI108419. PMID 932191
- [Background] Lumb MJ, Birdsey GM, Danpure CJ. Correction of an enzyme trafficking defect in hereditary kidney stone disease in vitro. Biochem J. 2003 Aug 15;374(Pt 1):79-87. doi: 10.1042/BJ20030371. PMID 12737622
- [Background] Lumb MJ, Danpure CJ. Functional synergism between the most common polymorphism in human alanine:glyoxylate aminotransferase and four of the most common disease-causing mutations. J Biol Chem. 2000 Nov 17;275(46):36415-22. doi: 10.1074/jbc.M006693200. PMID 10960483
- [Background] Monico CG, Rossetti S, Olson JB, Milliner DS. Pyridoxine effect in type I primary hyperoxaluria is associated with the most common mutant allele. Kidney Int. 2005 May;67(5):1704-9. doi: 10.1111/j.1523-1755.2005.00267.x. PMID 15840016
- [Background] Purdue PE, Takada Y, Danpure CJ. Identification of mutations associated with peroxisome-to-mitochondrion mistargeting of alanine/glyoxylate aminotransferase in primary hyperoxaluria type 1. J Cell Biol. 1990 Dec;111(6 Pt 1):2341-51. doi: 10.1083/jcb.111.6.2341. PMID 1703535
- [Background] Rantanen I, Nicander I, Jutila K, Ollmar S, Tenovuo J, Soderling E. Betaine reduces the irritating effect of sodium lauryl sulfate on human oral mucosa in vivo. Acta Odontol Scand. 2002 Oct;60(5):306-10. doi: 10.1080/00016350260248292. PMID 12418722
- [Background] Santana A, Salido E, Torres A, Shapiro LJ. Primary hyperoxaluria type 1 in the Canary Islands: a conformational disease due to I244T mutation in the P11L-containing alanine:glyoxylate aminotransferase. Proc Natl Acad Sci U S A. 2003 Jun 10;100(12):7277-82. doi: 10.1073/pnas.1131968100. Epub 2003 May 30. PMID 12777626
- [Background] Schwahn BC, Hafner D, Hohlfeld T, Balkenhol N, Laryea MD, Wendel U. Pharmacokinetics of oral betaine in healthy subjects and patients with homocystinuria. Br J Clin Pharmacol. 2003 Jan;55(1):6-13. doi: 10.1046/j.1365-2125.2003.01717.x. PMID 12534635
- [Background] Voziyan PA, Fisher MT. Polyols induce ATP-independent folding of GroEL-bound bacterial glutamine synthetase. Arch Biochem Biophys. 2002 Jan 15;397(2):293-7. doi: 10.1006/abbi.2001.2620. PMID 11795885
- [Background] Micromedex Healthcare Series (http://wwwmicromed.mayo.edu).
- [Background] Berlow S, Bachman RP, Berry GT, Donnell GN, Grix A, Levitsky LL, Hoganson G, Levy HL. Betaine therapy in homocystinemia. Brain Dysfunct 2:10-24, 1989.
- [Background] Smolin LA, Benevenga NJ, Berlow S. The use of betaine for the treatment of homocystinuria. J Pediatr. 1981 Sep;99(3):467-72. doi: 10.1016/s0022-3476(81)80352-6. No abstract available. PMID 7264811
- [Background] Holme E, Kjellman B, Ronge E. Betaine for treatment of homocystinuria caused by methylenetetrahydrofolate reductase deficiency. Arch Dis Child. 1989 Jul;64(7):1061-4. doi: 10.1136/adc.64.7.1061. PMID 2629632
- [Background] Wilcken DE, Wilcken B, Dudman NP, Tyrrell PA. Homocystinuria--the effects of betaine in the treatment of patients not responsive to pyridoxine. N Engl J Med. 1983 Aug 25;309(8):448-53. doi: 10.1056/NEJM198308253090802. PMID 6877313
- [Background] Dudman NP, Guo XW, Gordon RB, Dawson PA, Wilcken DE. Human homocysteine catabolism: three major pathways and their relevance to development of arterial occlusive disease. J Nutr. 1996 Apr;126(4 Suppl):1295S-300S. doi: 10.1093/jn/126.suppl_4.1295S. PMID 8642474
- [Background] McGregor DO, Dellow WJ, Robson RA, Lever M, George PM, Chambers ST. Betaine supplementation decreases post-methionine hyperhomocysteinemia in chronic renal failure. Kidney Int. 2002 Mar;61(3):1040-6. doi: 10.1046/j.1523-1755.2002.00199.x. PMID 11849459
- [Background] van Guldener C, Janssen MJ, de Meer K, Donker AJ, Stehouwer CD. Effect of folic acid and betaine on fasting and postmethionine-loading plasma homocysteine and methionine levels in chronic haemodialysis patients. J Intern Med. 1999 Feb;245(2):175-83. doi: 10.1046/j.1365-2796.1999.00430.x. PMID 10081520
- [Background] van Guldener C, Lambert J, ter Wee PM, Donker AJ, Stehouwer CD. Carotid artery stiffness in patients with end-stage renal disease: no effect of long-term homocysteine-lowering therapy. Clin Nephrol. 2000 Jan;53(1):33-41. PMID 10661480
- [Background] Matthews A, Johnson TN, Rostami-Hodjegan A, Chakrapani A, Wraith JE, Moat SJ, Bonham JR, Tucker GT. An indirect response model of homocysteine suppression by betaine: optimising the dosage regimen of betaine in homocystinuria. Br J Clin Pharmacol. 2002 Aug;54(2):140-6. doi: 10.1046/j.1365-2125.2002.01620.x. PMID 12207633
- [Background] Surtees R, Bowron A, Leonard J. Cerebrospinal fluid and plasma total homocysteine and related metabolites in children with cystathionine beta-synthase deficiency: the effect of treatment. Pediatr Res. 1997 Nov;42(5):577-82. doi: 10.1203/00006450-199711000-00004. PMID 9357926
- [Background] Wendel U, Bremer HJ. Betaine in the treatment of homocystinuria due to 5,10-methylenetetrahydrofolate reductase deficiency. Eur J Pediatr. 1984 Jun;142(2):147-50. doi: 10.1007/BF00445602. PMID 6381059
- [Background] Devlin AM, Hajipour L, Gholkar A, Fernandes H, Ramesh V, Morris AA. Cerebral edema associated with betaine treatment in classical homocystinuria. J Pediatr. 2004 Apr;144(4):545-8. doi: 10.1016/j.jpeds.2003.12.041. PMID 15069409
- [Background] Yaghmai R, Kashani AH, Geraghty MT, Okoh J, Pomper M, Tangerman A, Wagner C, Stabler SP, Allen RH, Mudd SH, Braverman N. Progressive cerebral edema associated with high methionine levels and betaine therapy in a patient with cystathionine beta-synthase (CBS) deficiency. Am J Med Genet. 2002 Feb 15;108(1):57-63. doi: 10.1002/ajmg.10186. PMID 11857551
- See also: Mayo Clinic Hyperoxaluria Center home page — http://www.mayoclinic.org/nephrology-rst/hyperoxaluriacenter.html
- See also: Mayo Clinic Hyperoxaluria Center (disease web page) — http://www.mayoclinic.org/hyperoxaluria/
- See also: Oxalosis and Hyperoxaluria Foundation — http://www.ohf.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic, Rochester between October 2006 and September 2008.
Pre-assignment Details: Fifteen subjects were enrolled, but 2 subjects withdrew prior to group assignment.
Groups:
- Betaine First, Then Placebo: Subjects received oral betaine 10 gm (subjects >10 yrs old) or 6 gm (subjects <10 yrs old) divided in two doses daily, for 2 months, followed by a 2 month washout period. Subjects then received oral lactose placebo divided in two doses daily, for 2 months.
- Placebo First, Then Betaine: Subjects received oral lactose placebo divided in two doses daily, for 2 months, followed by a 2 month washout period. Subjects then received oral betaine 10 gm (subjects >10 yrs old) or 6 gm (subjects <10 yrs old), divided in two doses daily, for 2 months.
Period: First Intervention
Arm/Group | Betaine First, Then Placebo | Placebo First, Then Betaine
Started | 6 | 7
Completed | 5 | 5
Not Completed | 1 | 2
Not completed — Subject non-compliant | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period of 2 Months
Arm/Group | Betaine First, Then Placebo | Placebo First, Then Betaine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Betaine First, Then Placebo | Placebo First, Then Betaine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive placebo first and betaine first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 20.1 [6 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13
Glomerular Filtration Rate (GFR) [Mean (Full Range); unit: ml/min/1.73 m^2] | 79 [39 to 134]
Number of Subjects on Concomitant Medications [Number; unit: participants] — Usual medications for primary hyperoxaluria were continued throughout the study. Subjects could have been prescribed more than one medication, so the sum of participants will be greater than the subject population.
  participants
    Vitamin B6 | 9
    Neutral Phosphate | 7
    Citrate | 3

OUTCOME MEASURES:

1. Primary Outcome: Urinary Oxalate Excretion
Description: The patients were randomly assigned oral betaine or placebo for 2 months, followed by a 2 month washout. Each patient then received the alternate study medication for 2 months.
  Urinary Oxalate Excretion was measured by oxalate oxidase. Two 24 hour urine collections were obtained at baseline, and during the eighth week of each study period.
Time Frame: baseline, 2 months, 6 months
Population: Per protocol analysis: 10 of 15 enrolled PHI subjects completed the study: 2 withdrew before initiation, 2 were noncompliant, in 1 symptoms led to withdrawal.
Measure: Mean (Standard Deviation); unit: umol/mg
Groups:
- Betaine: Subjects received oral betaine 10 gm (subjects >10 yrs old) or 6 gm (subjects <10 yrs old), divided in two doses daily, for 2 months.
- Placebo: Subjects received oral lactose placebo divided in two doses daily, for 2 months.
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 10 | 10
umol/mg | 1.43 (0.97) | 1.04 (0.71)
Statistical Analysis 1: Comparison: Betaine vs Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects will be followed for adverse events for the 6 months while on study.
Description: Subjects unable to tolerate the initial dose due to gastrointestinal symptoms will be offered a dose reduction of 3 - 5 g/day. Monitoring for symptoms and signs of cerebral edema will be 1) weekly telephone calls from the study coordinator with a list of questions re: increased intracranial pressure and 2) full eye exam before and after treatment.
Arm/Group | Betaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 11/13 | 8/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betaine (N=13) | Placebo (N=13)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 7 (7)
Diarrhea/loose stools (Gastrointestinal disorders) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Headache (General disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No